CLINICAL TRIAL: NCT07379437
Title: Effects and Mechanism of Haematococcus Pluvialis Astaxanthin on Inhibiting Brain Aging Through Improving Mitochondrial Function
Brief Title: Haematococcus Pluvialis Astaxanthin for Brain Aging
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Miao Chen, Doctoral Student, Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CNS-NCL2024-04
Record Dates: First submitted 2025-12-21; First posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Brain Aging

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo Group (Placebo Comparator): Placebo
  Interventions: Other: Placebo
- Low-Dose AST Group (Experimental): 6 mg/d Astaxanthin (Haematococcus pluvialis)
  Interventions: Dietary Supplement: Low-Dose AST
- High-Dose AST Group (Experimental): 12 mg/d Astaxanthin (Haematococcus pluvialis)
  Interventions: Dietary Supplement: High-Dose AST

INTERVENTIONS:
Dietary Supplement: Low-Dose AST — Low-Dose AST Group:6 mg/d Astaxanthin (Haematococcus pluvialis)
  Arms: Low-Dose AST Group
Dietary Supplement: High-Dose AST — High-Dose Group: 12 mg/d Astaxanthin (Haematococcus pluvialis)
  Arms: High-Dose AST Group
Other: Placebo — Placebo
  Arms: Placebo Group

SUMMARY:
We recruit community-dwelling older adults aged 50 and above for a 6-month intervention. Participants are divided into three groups:

Placebo Group, Low-Dose Group ( 6 mg/d Haematococcus pluvialis Astaxanthin), High-Dose Group (12 mg/d Haematococcus pluvialis Astaxanthin).

Peripheral blood samples and Other tests are collected at baseline, 3 months, and 6 months to measure mitochondrial function and oxidative stress levels.

Assessments include: 1.Cognitive & Neurophysiological Assessment: Using the MoCA (Montreal Cognitive Assessmentscale) and ERP (specifically P300) monitoring. 2.Brain Imaging: MRI (Magnetic resonance imaging) is used to analyze changes in brain function. 3.Metabolomics: A series of laboratory techniques are used to analyze routine metabolic indices, plasma astaxanthin, mitochondrial function, oxidative stress markers, and cognition-related neurobiomarkers.

DETAILED DESCRIPTION:
This study proposed to set the intervention doses at 6 mg/day and 12 mg/day, with an intervention period of 6 months. The intervention agent was Astaxanthin Capsules from Haematococcus pluvialis (containing 6 mg of astaxanthin per capsule) supplied by Astareal Corporation, Japan. The control group received placebo capsules identical to the intervention group in terms of color, shape, size, packaging, and quantity but devoid of astaxanthin. Prior to the experiment, random sampling was conducted on the intervention capsules to verify the effective content of astaxanthin, ensuring the accuracy of the intervention doses. During the intervention period, experimenters distributed the intervention and control capsules to the corresponding populations, along with a consumption record form. The dosage for each month was administered, and the capsule containers were collected at the end of each month. Daily text messages were sent to remind participants to take the capsules and check in, with compliance assessed based on the record form and check-in records.A self-designed questionnaire was used to conduct baseline surveys on the study subjects, covering demographic characteristics, lifestyle, and medical history. The demographic survey included gender, age, educational level, marital status, occupation, and housing conditions. Lifestyle factors were assessed through smoking, alcohol consumption, mental activity (e.g., reading, newspaper consumption, computer use, television viewing), physical activity, household chores, and dietary supplement use. Past medical history encompassed current illnesses, prior diseases, family genetic history, duration of illness, and medication regimens. Physical examinations were performed by community health center physicians, measuring routine parameters such as height, weight, waist circumference, and blood pressure, with calculation of body mass index (BMI).The dietary questionnaire designed by the research team was administered through face-to-face interviews by specially trained investigators.Cognitive function was measured before intervention (baseline), at 3 months of intervention, and at the end of intervention (6 months of intervention), including the following tests: 1) Tracking the changes in the brain's neural electrophysiology during cognitive processes using event-related potential (ERP) P300.2) The Montreal Cognitive Assessment (MoCA) was used to evaluate the cognitive function of the subjects.The Siemens Trio 3T MRI system was used to acquire imaging data, including T1-weighted structural and resting-state functional scans as well as T2w-FLAIR images.Fasting peripheral blood samples were collected at three time points (pre-intervention, 3 months, and 6 months), and after processing, underwent comprehensive laboratory analyses including routine metabolic panels, plasma astaxanthin, mitochondrial function, oxidative stress markers, and cognition-related neurobiomarkers.

ELIGIBILITY:
Inclusion Criteria:

Cognitive functionally normal elderly individuals aged 50 years or older with baseline MoCA scores near the borderline for mild cognitive impairment (MCI); subjects reporting age-related forgetfulness; community-dwelling residents who can cooperate with the research team to complete the intervention study.

Exclusion Criteria:

Individuals with hearing or language expression impairments that hinder communication; those with severe cardiovascular, cerebrovascular, hepatic, renal, or other organ diseases, or malignant tumors; individuals who have been taking astaxanthin or other antioxidant dietary supplements within the past month; those who have recently used medications that may affect neurological function; and individuals who are unable to undergo cognitive function assessment or refuse to sign an informed consent form.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2026-05-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Montreal Cognitive Assessment, MoCA | From enrollment to the end of treatment at 6 months
  The cognitive domains assessed included attention and concentration, executive function, memory, language, visual structural skills, abstract thinking, as well as calculation and orientation. The total score of the scale was 30 points.A total score of 26 or above is considered normal (as there is no current Chinese reliability and validity analysis, so the original foreign language threshold values can be temporarily referred to); a score of 19 to 25 indicates that there is a possibility of mild cognitive impairment (MCI); if the score is 19 to 22 and there is also some difficulty in daily life/activities, it usually means that the person has progressed from MCI to dementia; those with a score below 19 can clearly be diagnosed as having dementia.
Neurophysiology changes | From enrollment to the end of treatment at 6 months
  The event-related potential (ERP) P300 was used to track the changes of the brain's neural electrophysiology during the cognitive process.Patients with cognitive decline and Alzheimer's disease show an extended P300 latency period.

SECONDARY OUTCOMES:
MRI（Magnetic resonance imaging） | From enrollment to the end of treatment at 6 months
  The Siemens Trio 3T MRI system was used to acquire imaging data, including T1-weighted structural and resting-state functional scans as well as T2w-FLAIR images.The common local brain structural changes associated with cognitive decline are the atrophy of the hippocampus and the entorhinal cortex.

CONTACTS AND LOCATIONS:
Overall Officials: Linhong Yuan, Doctor, Principal Investigator — Capital Medical University

IPD SHARING:
Plan to Share IPD: No